CLINICAL TRIAL: NCT02357563
Title: Ulipristal Acetate Versus GnRH Analogue for Myometrial Preservation in Patients With Submucosal Uterine Leiomyoma G2
Brief Title: Ulipristal Acetate Versus GnRH Analogue and Myometrial Preservation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPA myometrial
Record Dates: First submitted 2015-02-02; First posted 2015-02-06 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Fibroid
Keywords: fibroid; GnRH analogue; ulipristal acetate
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; Leuprolide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulipristal acetate (Experimental): Women will be treated with an oral dose of ulipristal acetate 5 mg/day for 2 courses of 3 months each
  Interventions: Drug: ulipristal acetate
- Leuprolile acetate (Active Comparator): Women will be treated with an injection IM on leuprolide acetate 11,25 in the luteal phase repeated 3 months later
  Interventions: Drug: Leuprolide acetate

INTERVENTIONS:
Drug: ulipristal acetate — 5 mg/day will be administered starting from day 1 of the cycle and up to three months later for two courses, with an interval between the courses of 1 month
  Other Names: Esmya
  Arms: Ulipristal acetate
Drug: Leuprolide acetate — One dose of 11.25 GnRH analogue depot will be administered in the luteal phase of the menstrual cycle (days 21-24) and repeated 3 months later
  Other Names: Enantone 11.25
  Arms: Leuprolile acetate

SUMMARY:
Submucosal fibroid grow inside the uterine cavity and are associated with menorrhagia, abnormal uterine bleeding (AUB) and infertility. Type II (G2) fibroids often require more surgeries due to their particular position in the myometrium. Surgery, moreover, should always be tailored, particularly in patients wishing to conceive, to preserve the integrity of the myometrium. Preoperative use of GnRH agonist appears to be relevant and beneficial in patients with submucous fibroids, but are associated with several side effects. the eighty percent of patients treated by UPA showed a clinically meaningful reduction of more than 25% in fibroid volume, and 50% of patients a reduction of 50%. fibroid volume reduction appeared to be maintained for 6 months after the end of UPA treatment

DETAILED DESCRIPTION:
Uterine leiomyoma is the most common benign tumor of the female genital tract. Submucosal fibroid are about 10% of all uterine myoma. They grow inside the uterine cavity and are usually associated with menorrhagia, abnormal uterine bleeding (AUB) and infertility. According to the degree of myometrial penetration, the European Society for Gynaecological Endoscopy (ESGE) classified submucosal myomas in Type 0 (G0, totally intracavitary fibroids), Type I (G1, <50% myometral penetration), or Type II (G2, >50% myometral penetration).

Hysteroscopic removal of submucosal myomas improves menorrhagia and AUB but can be challenging in women with Type II (G2) fibroids, since they often require more and more surgeries due to their particular position in the context of myometrium. Surgery, moreover, should always be tailored, particularly in patients wishing to conceive, to preserve the integrity of the myometrium. In this particular population, indeed, the possibility of avoiding any kind of uterine surgery should always be exploited. Up to now, hysteroscopic resection of submucosal fibroids is considered the gold standard for symptomatic patients, since no medication has been able to restore uterine cavity in a permanent manner. In this setting, use of a GnRH agonist before surgery is still a matter of debate, but literature reports that preoperative use of GnRH agonist appears to be relevant and beneficial in patients with submucous fibroids. Benefits include a resolution of preoperative anemia, a decrease in fibroid size, a reduction of endometrial thickness and vascularization with subsequently improved visibility and reduced fluid absorption, and the possibility of surgical scheduling.

Conversely, this preoperative treatment is associated with some side effects such as hot flushes and postinjection endometrial bleeding due to the flare-up effect.

Data on SPRM showed that eighty percent of patients treated by UPA showed a clinically meaningful reduction of more than 25% in fibroid volume, and 50% of patients a reduction of 50%. In the subpopulation of patients not undergoing surgery, fibroid volume reduction appeared to be maintained for 6 months after the end of UPA treatment.

This was in contrast to patients receiving a GnRH agonist, in whom fibroids began to regrow 1 to 3 months after the last dose, reaching their baseline size after 6 months.

No sub-analysis have been conducted on submucosal fibroids, but is of interest to underline that, when myomas regress so much that they no longer distort the uterine cavity, surgery may not be required. This could represent a safe way to avoid surgery in patients with G2 fibroids desiring pregnancy.

ELIGIBILITY:
Inclusion Criteria:

G2 submucosal leiomyoma <3 cm, symptoms of menomethrorragia, menstrual disorder, infertility, pelvic pain

Exclusion Criteria:

submucosal leyomyoma other than G2 or greater than 3 cm, intramural or subserosal leiomyomas endometrial hyperplasia with atypia history of uterine surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of restored uterine cavity 1 year after enrollment | 1 year after treatment
  To compare the proportion of patients, treated by UPA or by GnRh-a, with uterine cavity no longer distorted by their submucous myoma

SECONDARY OUTCOMES:
Time to pregnancy | from the end of treatment to the obtainance of pregnancy
  to compare time to pregnancy in patients treated with Ulipristal Acetate and GnRH-a
Live birth rate | A the time of delivery
  to compare live birth rate in patients treated with Ulipristal Acetate and GnRH-a
Proportion of patients needing surgery after UPA or GnRH-a | 24 weeks after the first dose of drugs
  to compare need for surgery in patients treated with Ulipristal Acetate and GnRH-a.

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD,PhD, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, MD, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, Catanzaro, Italy